CLINICAL TRIAL: NCT06161740
Title: Effect of Low-intensity Aerobic Training Associated With Global Muscle Strengthening in Post-COVID-19 Individuals
Brief Title: Low-intensity Aerobic Training Associated With Global Muscle Strengthening in Post-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUPAC
Record Dates: First submitted 2023-12-05; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Rehabilitation; Physiotherapy; Endurance training; Medical Research Council; Quality of Life
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle strengthening group MSG (Active Comparator): It was based on exercises for strengthening the hip adductor muscles associated with a bridge using a small exercise ball (two sets of 15 repetitions with seven seconds in isometry), strengthening the hamstrings with ankle weights in prone position, bilateral hip flexor strengthening in supine position with ankle weights, bilateral shoulder flexor strengthening with dumbbells, bilateral shoulder extensor strengthening with dumbbells, bilateral shoulder abductor strengthening with dumbbells, and bilateral serratus anterior muscle strengthening with dumbbells (all exercises, except the first, performed in three sets of 10 repetitions). Considering a 15-second interval between repetitions and a one-minute break between sets, totaling 30 minutes. The progression of each patient occurred through load progression.
  Interventions: Procedure: muscle strengthening
- Muscle strengthening associated with aerobic training group (MSGA) (Experimental): It initially consisted of a five-minute warm-up, divided into two minutes of stationary marching and three minutes of jumping jacks. Subsequently, patients were instructed to climb up and down ramps, ascend and descend stairs, walk on a flat surface, and use a cycle ergometer (each task performed for five minutes). For the recovery phase, bilateral stretching of the hamstrings, rectus femoris, triceps brachii, pectoralis major, sternocleidomastoid, and scalene muscles was performed, each lasting 30 seconds per muscle. The proposed protocol was associated with the anaerobic training described in the GF (muscle strengthening group).
  Interventions: Procedure: muscle strengthening

INTERVENTIONS:
Procedure: muscle strengthening — The study involved adults aged 18 to 59 diagnosed with COVID-19 in the past year, experiencing mild or moderate symptoms, dyspnea, and either sedentary or engaging in physical exercise at least twice a week. Excluded were those with certain medical conditions. The participants were divided into two groups: one focused on global muscle strengthening (GF), and the other on low-intensity aerobic training with global muscle strengthening (GAF). The study assessed various parameters, including BMI, quality of life, aerobic capacity, dyspnea, and muscle strength. The sessions varied in duration and intensity. Volunteers were recruited from a clinic in Ubá-MG and randomly assigned to groups. The study aimed to evaluate the impact of the interventions on post-COVID-19 recovery.
  Other Names: aerobic exercises

SUMMARY:
The study called "Effect of low-intensity aerobic training associated with global muscle strengthening in post-COVID-19 individuals" wants to check if doing easy workouts and strengthening muscles can make breathing problems better for adults who had COVID-19.

The participant has been apprised that potential benefits may be derived from the research, including the reception of treatment for pertinent complaints meeting the study's inclusion criteria. Conversely, they have also been briefed on possible discomforts and risks associated with the study, such as the exposure of their image to the therapist administering the treatment.

The participant acknowledges that their privacy will be upheld, ensuring the confidentiality of personal information, including their name or any other identifying data. It has been communicated that the participant reserves the right to decline participation in the study or withdraw consent at any point without the obligation to provide justification. Moreover, they are assured that opting out of the study will not result in any adverse consequences.

DETAILED DESCRIPTION:
Patients of both genders aged 18 to 59 years were included in the study. They had been diagnosed with COVID-19 in the past year, experienced mild or moderate symptoms, had shortness of breath, were either sedentary or engaged in physical exercise at least twice a week, and agreed to sign the Informed Consent Form. Excluded from the study were individuals hospitalized due to COVID-19, those diagnosed with chronic lung diseases, smokers, those who had undergone prior physiotherapeutic treatment for post-COVID-19 syndrome, individuals with a history of lower limb surgeries or fractures (within the last six months), BMI over 30 kg/m², and those with neurological, cognitive, or cardiac impairments.

The sample, selected for convenience, was divided into two distinct groups: the global muscle strengthening group (GF) and the low-intensity aerobic training associated with global muscle strengthening group (GAF). The GF comprised eight volunteers, while the GAF had nine, totaling eight sessions with a frequency of two interventions per week, lasting 30 minutes each for the GF and 60 minutes each for the GAF. Two assessments were conducted: one at admission and another at the end of the treatment.

Participants were recruited at the Dr. Cícero Brandon School Clinic of Faculty President Antônio Carlos in Ubá city, state of Minas Gerais, with authorization for data collection and infrastructure use signed by the study researchers and supervisor. Volunteers were assessed during the first session to ensure compliance with inclusion and exclusion criteria outlined in the medical history form. They were informed about the entire procedure and study objectives and subsequently guided to sign the Informed Consent Form, following Resolution 466/2012 of the National Health Council.

Body Mass Index (BMI) calculation was done using a Multilaser digital scale and a two-meter measuring tape. Quality of life was assessed using the abbreviated version of the WHOQOL-100, the WHOQOL-bref, consisting of 26 questions related to general quality of life, satisfaction with one's health, and domains of physical, psychological, social relationships, and the environment.

Aerobic capacity was evaluated through the Six-Minute Walk Test (6MWT), performed on a flat, obstacle-free 30-meter track. The objective was to analyze the farthest distance a patient could walk in six minutes without running, with the option to stop at any time without interrupting the timing. Standardized encouragement phrases were used every minute during the test.

The Medical Research Council (MRC) Dyspnea Scale was used to categorize the degree of dyspnea, with patients choosing an item corresponding to the proportion of limitation caused by dyspnea in their daily activities. Muscle strength measurement was conducted for each volunteer using a validated digital scale in the quadriceps (90° knee flexion), hamstrings (90° knee flexion), biceps brachii (90° elbow flexion), triceps brachii (anatomical position), and deltoid (midportion, 30° shoulder abduction).

Blood pressure, heart rate, and oxygen saturation were measured at the beginning and end of each session using a premium brand sphygmomanometer and stethoscope, a G-tech pulse oximeter, and assessed throughout the session. Difficulty levels in performing proposed activities, considering peripheral musculature, were queried using the Borg Scale.

The GF group focused on exercises for strengthening hip adductor muscles associated with bridge exercises using a small exercise ball, hamstring strengthening with ankle weights in prone position, bilateral hip flexor strengthening in supine position with ankle weights, bilateral shoulder flexor strengthening with dumbbells, bilateral shoulder extensor strengthening with dumbbells, bilateral shoulder abductor strengthening with dumbbells, and bilateral serratus anterior muscle strengthening with dumbbells (all exercises except the first in three sets of 10 repetitions). Progression was based on each patient's development.

The GAF protocol initially involved a five-minute warm-up, consisting of two minutes of stationary marching and three minutes of jumping jacks. Patients were then instructed to climb up and down ramps, ascend and descend stairs, walk on a flat surface, and use a cycle ergometer (each task performed for five minutes). For the recovery phase, bilateral stretching of hamstrings, rectus femoris, triceps brachii, pectoralis major, sternocleidomastoid, and scalene muscles was performed, each lasting 30 seconds. This protocol was associated with the anaerobic training described in the GF.

Volunteers were allocated to two groups using a simple random sampling method with two blocks. Results were placed in sealed envelopes, concealing the patient allocation sequence from the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aged 18 to 59 diagnosed with COVID-19 in the past year
* Patients experienced mild or moderate symptoms
* Sedentary or engaged in physical exercise at least twice a week

Exclusion Criteria:

* Patients hospitalized due to COVID-19 diagnosed with chronic lung diseases
* Patients underwent prior physiotherapeutic treatment for post-COVID-19 syndrome
* History of surgeries or fractures in the lower limbs (within the last six months)
* BMI over 30 kg/m²
* Patients with neurological, cognitive, or cardiac impairments

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of life score | WHOQOL-bref questionnaire score was calculated before and after intervention, with a follow up of two months.
  The low-intensity aerobic training associated with overall muscle strengthening will promote quality of life.

SECONDARY OUTCOMES:
Dyspnea score | MRC scale score was assessed before and after intervention, with a follow up of two months
  The low-intensity aerobic training associated with overall muscle strengthening will promote an effect, reducing dynapenia and dyspnea in adults post-COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Hebert Olímpio Júnior, Divinésia, Brasil (+55), Brazil

IPD SHARING:
Plan to Share IPD: No